CLINICAL TRIAL: NCT00978718
Title: Phase III Trial of Selenium for Prostate Cancer Prevention
Brief Title: Selenium in Preventing Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 01-0506-01; R01CA077789 (NIH); P30CA023074 (NIH); UARIZ-99-0045-01, (Other: CDR0000654651)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenium

ARMS (3):
- Arm I (Placebo Comparator): Patients receive oral placebo daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.
  Interventions: Other: placebo
- Arm II: 200 μg selenium (Se) as high-Se Baker's yeast daily (Experimental): Patients receive 200 μg of oral selenium (Se) as high-Se Baker's yeast daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.
  Interventions: Dietary Supplement: selenium
- Arm III: 400 μg Se as high-Se baker's yeast daily (Experimental): Patients receive 400 μg of oral Se as high-Se baker's yeast daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.
  Interventions: Dietary Supplement: high-selenium baker's yeast

INTERVENTIONS:
Dietary Supplement: high-selenium baker's yeast — Given orally
  Other Names: selenium
  Arms: Arm III: 400 μg Se as high-Se baker's yeast daily
Dietary Supplement: selenium — Given orally
  Arms: Arm II: 200 μg selenium (Se) as high-Se Baker's yeast daily
Other: placebo — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Selenium supplements may stop or delay the development of prostate cancer in patients at high risk of prostate cancer. It is not yet known which dose of selenium may be more effective in preventing prostate cancer.

PURPOSE: This randomized phase III trial is studying how well selenium works in preventing prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether selenium (Se) supplementation decreases the incidence of prostate cancer.
* To determine whether Se supplementation inhibits the biochemical progression of prostate cancer.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral placebo daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.
* Arm II: Patients receive 200 μg of oral selenium (Se) as high-Se Baker's yeast daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.
* Arm III: Patients receive 400 μg of oral Se as high-Se baker's yeast daily. Treatment continues for up to 57 months in the absence of unacceptable toxicity or diagnosis of prostate cancer.

Blood samples are collected at baseline, at randomization, and then semi-annually for laboratory and other testing. Tissue samples may also be collected for biomarker analysis. Patients complete an initial questionnaire and urological-symptoms questionnaire at baseline, a follow-up questionnaire after randomization (to capture new illness, medications, and toxicity symptoms during the 30-day run-in period; a urological-symptoms questionnaire; a food-frequency questionnaire; and a mood questionnaire). Patients then undergo questionnaires semi-annually, including vital status, tablet compliance, nutrition, mood, new illnesses or medications, and any incidence of cancer or family history of cancer).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical indicators consistent with the community standards of medical care that would justify a biopsy of the prostate for the diagnosis of cancer, including ≥ 1 of the following:

  * PSA level above the absolute value of 4 ng/mL or above a published age-ethnic adjusted PSA level appropriate for the community
  * Rising PSA that should represent a clinically significant PSA velocity (e.g., an estimated annual change in the PSA velocity ≥ 0.75 ng/mL)
  * Abnormal digital rectal examination of the prostate that identifies a clinically significant change in the prostate (e.g., a prostate nodule or a change in the firmness of the prostate)
  * Documentation of the clinical assessment that justified the prostate biopsy that allows classification of the patient to high-risk groups
* Prostate biopsy negative for cancer within the past 12 months
* Prostate biopsy negative for high-grade prostatic intraepithelial neoplasia (PIN)

  * PIN allowed provided it is grade 1

PATIENT CHARACTERISTICS:

* Creatinine < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* SGOT and SGPT < 2 times ULN
* Alkaline phosphatase < 2 times ULN
* No history of a prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell carcinoma
  * Adequately treated (i.e., complete surgical removal with negative margins) stage I cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy or radiotherapy
* At least 90 days since prior and no other concurrent selenium > 55 μg/day as a dietary supplement (including multivitamin supplements)
* More than 30 days since prior and no concurrent participation in any other clinical trial involving a medical, surgical, nutritional, or life-style intervention (e.g., dietary modifications, exercise)

Max Age: 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2001-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-proven prostate cancer

SECONDARY OUTCOMES:
Rate of rise in serum PSA levels
Evidence of prostate cancer progression as assessed by levels of the serum markers alkaline phosphatase and Chromogranin A

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R. Ahmann, MD, Principal Investigator — University of Arizona